CLINICAL TRIAL: NCT02969421
Title: A Randomized Controlled Study of Patient Pain Perception With Tenaculum Placement During In-office Procedures
Brief Title: Pain Perception With Tenaculum Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00078232
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow Tenaculum Placement (Active Comparator): This group will have their tenaculum placed using the slow method
  Interventions: Other: Slow Tenaculum Placement of tenaculum
- Cough Method (Active Comparator): This group will have their tenaculum placed using the cough method
  Interventions: Other: Cough method for placement of tenaculum

INTERVENTIONS:
Other: Cough method for placement of tenaculum — The intervention in this arm is the placement of tenaculum via cough method
  Arms: Cough Method
Other: Slow Tenaculum Placement of tenaculum — The intervention in this arm is the placement of tenaculum via slow method
  Arms: Slow Tenaculum Placement

SUMMARY:
Randomized controlled trial that compares methods of tenaculum placement during intrauterine device insertion and their effect on pain. The two methods being compared are slow tenaculum placement versus tenaculum placement at time of cough. Subjects will be asked to rate their pain using visual analog scale. Primary outcome measured is pain at time of tenaculum placement. Secondary outcomes are overall pain with intrauterine device insertion and provider satisfaction with tenaculum placement.

DETAILED DESCRIPTION:
The two commonly described strategies for tenaculum placement, slow versus having the patient cough while the tenaculum is placed are utilized by providers based on preference and/or their previous training. There is no published study that compares these methods to one another. The investigators aim to compare these strategies, slow tenaculum placement versus the cough method, and their effects on pain at time of placement. 96 subjects will be randomized to each method. The subject will be asked to rate their pain using a 100-mm visual analog scale after speculum placement, after tenaculum is placed, and after completion of the procedure. The provider will be asked to rate their satisfaction with tenaculum placement on a Likert-type 5 point satisfaction scale. 1: not at all satisfied, 2: slightly satisfied, 3: moderately satisfied, 4: very satisfied, 5: extremely satisfied. All data to be collected using REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 years and older
* Undergoing intrauterine device placement
* English or Spanish speaking

Exclusion Criteria:

* Primary language other than English or Spanish

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

REFERENCES:
- [Derived] Lambert T, Truong T, Gray B. Pain perception with cervical tenaculum placement during intrauterine device insertion: a randomised controlled trial. BMJ Sex Reprod Health. 2020 Apr;46(2):126-131. doi: 10.1136/bmjsrh-2019-200376. Epub 2019 Oct 30. PMID 31666302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Slow Tenaculum Placement | Cough Method
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Slow Tenaculum Placement | Cough Method | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [21 to 31] | 28 [18 to 42] | 26 [22.2 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 9 | 22
  White | 13 | 19 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12
Number of Participants with Parity >=1 [Count of Participants; unit: Participants] | 14 | 19 | 33
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 26.4 [23 to 36.5] | 24.8 [22 to 38.1] | 26.1 [22.2 to 37.6]

OUTCOME MEASURES:

1. Primary Outcome: Pain With Tenaculum Placement
Description: Measured using 100-mm visual analog scale. Minimum value 0 meaning no pain and maximum value of 100 meaning worst imaginable pain.
Time Frame: Directly after tenaculum placement
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Slow Tenaculum Placement | Cough Method
Number analyzed (Participants) | 33 | 33
units on a scale | 44 [21 to 63] | 32 [19 to 54]

2. Secondary Outcome: Overall Pain With Intrauterine Device Insertion
Description: as for outcome 1
Time Frame: Directly after intrauterine device is placed
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Slow Tenaculum Placement | Cough Method
Number analyzed (Participants) | 33 | 33
units on a scale | 62 [48 to 84] | 54 [32 to 71]

3. Secondary Outcome: Provider Satisfaction With Tenaculum Placement
Description: Measured using Likert-type 5 point satisfaction scale dichotomized to optimal (Likert score = 4 or 5) vs suboptimal (Likert score = 1, 2, 3). Reported is the number of participants with optimal grasp.
Time Frame: Directly after tenaculum is placed
Measure: Count of Participants; unit: Participants
Arm/Group | Slow Tenaculum Placement | Cough Method
Number analyzed (Participants) | 33 | 33
Participants | 26 | 27

ADVERSE EVENTS:
Time Frame: 10 - 15 minutes of patient contact during and immediately after IUD insertion.
Arm/Group | Slow Tenaculum Placement | Cough Method
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

LIMITATIONS AND CAVEATS:
1. Non-blinded study
2. No gold standard for pain analysis
3. Lack of accountability for confounder of anxiety/use of anxiolytics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT02969421/Prot_SAP_000.pdf